CLINICAL TRIAL: NCT01482585
Title: Prospective Study of Early-stage Lung Adenocarcinoma for Early Detection and Effective Treatment Strategy
Brief Title: Study of Early-stage Lung Adenocarcinoma for Early Detection and Effective Treatment Strategy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Korean Foundation for Cancer Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: SMC 2011-09-083
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Lung Adenocarcinoma
Keywords: lung adenocarcinoma; prognosis; tumor aggressiveness; imaging biomarker; genetic biomarker
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; DNA Copy Number Variations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung tissue, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- early stage lung adenocarcinoma
  Interventions: Other: CT, PET, copy number alteration

INTERVENTIONS:
Other: CT, PET, copy number alteration — Duel-energy CT, PET, copy number alteration

SUMMARY:
to determine the values of imaging and genetic biomarkers for prediction of tumor aggressiveness and prognosis in patient with early stage lung adenocarcinoma to Identify unique copy number alteration in patient with early stage lung adenocarcinoma to evaluate the long-term change of ground-glass nodule combined with lung adenocarcinoma to suggest a guideline for planning an appropriate follow-up examination and management

ELIGIBILITY:
Inclusion Criteria:

* A. Clinically and radiologically suspected lung adenocarcinoma
* B. Newly-diagnosed Stage I or II from the clinical work up including PET/CT
* C. Performance status of 0 to 1 on the ECOG scale
* D. Age 20 years or older
* E. Able to tolerable DECT imaging required by protocol
* F. Able to give study-specific informed consent

Exclusion Criteria:

* A. Prior malignancy
* B. planning of Definitive RTx 나 neoadjuvant CCRTx
* C. Poor cardiopulmonary reserve

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with stage I or II lung adenocarcinoma who plans curative operation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of tumor aggressiveness | five years

SECONDARY OUTCOMES:
prognosis of early stage lung adenocarcinoma following operation | five years

CONTACTS AND LOCATIONS:
Overall Officials: Young Mog Shim, Dr., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea